CLINICAL TRIAL: NCT04067193
Title: Usability Study of PARADE CONNECT Shoes, a Device to Detect Falls in Old People
Brief Title: E-vone® Use Detect Falls Among hOspitalized Patients in geRiAtric Medicine
Acronym: EDORA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2019/49
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-09

CONDITIONS: Patients Hospitalised in Geriatrics
Keywords: old people; fall; elderly; fall detection; usability; satisfaction; ergonomy; shoes
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- old geriatric inpatients: usability assessment after 24 to 72 hours of possible use of the device (PARADE CONNECT shoes)
  Interventions: Other: usability survey
- unformal caregivers: usability assessment after 24 to 72 hours of possible use of the device (PARADE CONNECT shoes) by their relative
  Interventions: Other: usability survey
- professional caregivers: usability assessment after the possible use of the device (PARADE CONNECT shoes) by 40 hospitalzed old patients in the geriatrics ward
  Interventions: Other: usability survey

INTERVENTIONS:
Other: usability survey — usability survey composed of subpart: System Usability Scale, questions about ergonomic, questions about design, question about global satisfaction.

SUMMARY:
This study evaluates the usability of a new remote warning system for fall in old people. This system is integrated in a shoe. Patients hospitalized in a geriatric ward but also their informal and professional caregivers will assess the usability of the device using a structured survey.

DETAILED DESCRIPTION:
Falls are a major health concerned because of their frequency and severity. It is estimated that 30% of people over 65 years old and 50% of those over 85 years old fall at least once a year. Falls are also one of the main factors of morbidity, mortality and early institutionalization for old people.

Preventive measures have been implemented to limit the recurrence of falls. Most of these preventive measures are secondary and tertiary prevention programs, such as MultiFactorial Interventions (MFIs). Home-based programs are under evaluation, but evidences of their effectiveness are currently controversial. Effects of prevention programs for in and outpatients remain modest. The objectives of these interventions are to decrease the frequency of falls but also to decrease the severity of falls.

The severity of falls is due to their physical complications (found in 50 to 55% of cases), their psychological complications (40%) but it is also reflected by the subsequent hospitalizations (20%), the acceleration of dependency (50%) and the institutionalizations (40%). Falls are complicated by death in 5% of cases.

In addition, the literature on fall complications is profuse. One of these complications is the hip fracture. Hip fracture is the main cause of mortality and loss of autonomy due to falls. However, in a previous study conducted by Bloch et al. in 2009 at Cochin Hospital, several indirect evidences tended to show that mortality from falls was related to the metabolic disorders linked to the extended stay on the ground, rather than to immediate traumatic consequences. As metabolic disorders reflects the time needed to be rescued, this article highlights the importance of using early warning systems to reduce the occurrence of such complications in old frail patients living alone, and unable to get up alone from the ground.

The most commonly used warning tools are remote assistance systems (necklace or bracelet) with a button to push in case of a fall. In the study conducted by Flemming et al. in 2008, when these systems are activated, the great majority of fallers are back on their feet within one hour after the alert. Nevertheless, of 143 old people living alone and unable to get up alone from the ground, only 28 were using a warning system. The reasons for non-use are as follows: the person does not have a warning remote assistance systems, the person owns a warning remote assistance systems but was not wearing it at the time of the fall, the person was wearing a warning remote assistance systems but was forgetting (or was in difficulty) to use it.

Many research projects on fall warning and detection systems have been initiated. In the 2018 meta-analysis by Nguyen et al., fall detection systems are divided into 2 groups: a pre and a post-fall group. In the latter group, the detection systems were mainly using 3D accelerators, gyroscopes, magnetometers or smartphones with the above-mentioned devices. However, to date, there is no reliable detection system on the market because some obstacles remain. These obstacles are concerning technology but also usability. Concerning technological issue, one of the problems remains the ability of devices to detect low kinetic falls, which is common in the elderly. Concerning usability, questions are for example the problem of the voluntary activation by the user of the most common devices, or the absence of wearing the device during numerous falls.

PARADE CONNECT would remove some of the usability obstacle typically associated with remote warning systems. Indeed, the system is activated independently of the will, cognitive state and consciousness of its user. The warning system is integrated into a shoe usually worn by the old people, with probably a less stigmatizing character of aging and loss of independence. This is why it seems important to us, as a first step, to evaluate its acceptability and usability by patients.

ELIGIBILITY:
Inclusion criteria:

* Patients :

  * Aged 65 years old and over
  * To be hospitalised in geriatric medicine department of Angers University Hospital
* Unformal caregivers :

  * Family members or relatives
  * Age 18 years and over
* Professional caregivers:

  * geriatric medicine department's staff of Angers University Hospital
  * aged of 18 years and over

Exclusion criteria:

* Patients :

  * To have motor disability or walking contraindications
  * To be under legal protection
* Refusal of participating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients are recruited during their hospitalisation in geriatric medicine. Relatives / unformal caregivers are recruited during the hospitalisation of patients in geriatric medicine. Professionnal caregivers are recruited in the acute care geriatric unit.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-10-30 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-05-03 (Estimated)

PRIMARY OUTCOMES:
Usability of the PARADE CONNECT shoes: Average of the usability scores | within 24 hours after removal of the device
  Average of the usability scores. Usability score is calculated using the responses to the validated System Usability Scale (SUS). An average score equal or over 70/100 will be considered as satisfying.

SECONDARY OUTCOMES:
Satisfaction of the PARADE CONNECT shoes: recommendation scale | within 24 hours after removal of the device
  Average recommendation score. Satisfaction score is calculated using the responses to the recommendation scale. This scale is a ten point's scale from 0 (I don't recommend at all) to 10 (I fully recommend). An average score greater than 5/10 would be acceptable, a score greater than or equal to 7/10 would be satisfactory.
Ergonomic of the PARADE CONNECT shoes | within 24 hours after removal of the device
  Average ergonomics score: The ergonomics score is a composite score based on the average of the answers to five ergonomics questions on a four-level Likert scale. The Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree). The average score is reported on ten. An average score greater than 5/10 would be acceptable, a score greater than or equal to 7/10 would be satisfactory.
Preferred shape for the PARADE CONNECT shoes | within 24 hours after removal of the device
  Three shape of shoes will be presented. Each participant will be asked about his preferred shape of shoes. The prefered shape will be the most choose shapenof shoes.
Acceptability of the PARADE CONNECT shoes: Average acceptability score | within 24 hours after removal of the device
  Average acceptability score: The acceptability score is assessed using a closed question. The response is based on a four-level Likert scale. The Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree). The average score is reported on ten. An average score greater than 5/10 would be acceptable, a score greater than or equal to 7/10 would be satisfactory.

CONTACTS AND LOCATIONS:
Overall Officials: Cédric Annweiler, MD, PhD, Principal Investigator — Angers University Hospital
Locations (1):
- Angers University Hospital, Angers, France